CLINICAL TRIAL: NCT06067347
Title: Integration of Machine Learning and Genomics to Predict Outcomes for Newly Diagnosed, Relapsed and Refractory Mature T-cell and NK/T-cell Lymphomas: a Global Study of the PETAL Consortium
Brief Title: A Global Study of the PETAL Consortium
Acronym: PETAL
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Salvia Jain, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 23-212
Record Dates: First submitted 2023-09-05; First posted 2023-10-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: T-Cell and NK-Cell Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — After centralized review of the archived FFPE lymphoma specimen and immunostains obtained at diagnosis, the pathology investigator at each participating institution will retain a Hematoxylin and Eosin (H&E) slide and send up to 20 de-identified unstained slides representative of the tumor to our genomics partner. These slides will undergo NGS, including bulk RNA-seq and WES. Where feasible, DNA extracted from mononuclear cells and saliva will also be sent for NGS as a germline control. Following quality control (QC) review, we will perform NGS and analysis, then share the raw data and results with the participating investigator from the institution that enrolled the research participant.
  We anticipate participation and enrollment from up to 20 global sites in this consortium.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Massachusetts General Hospital, Boston, USA: Participating investigators at various institutions will perform weekly review of their new patients with PTCL (newly diagnosed or relapsed/refractory) on the outpatient and inpatient clinical services with their clinical research teams to identify potential subjects for enrollment based on the above inclusion/exclusion criteria. Expected enrollment is anticipated to be up to 50 patients per site per year.

SUMMARY:
The goal of this observational study is to correlate molecular alterations with outcomes including overall survival (OS), progression-free survival (PFS), response rates for patients with a new diagnosis, primary refractory or relapse, of mature T-cell and NK-cell neoplasms (TNKL). We hypothesize that machine learning can be leveraged to uncover distinct genetic vulnerabilities that underlie treatment response and resistance for patients with TNKL, thus moving towards personalized treatment solutions.

DETAILED DESCRIPTION:
This study is a prospective, longitudinal observational study of patients with newly diagnosed or relapsed/refractory T-cell and NK-cell neoplasms, conducted across multiple participating institutions globally. Patients will be enrolled during their initial visit as new patients and will be followed for up to four years through the course of their clinical management. Data for routine demographics, baseline clinical features, including pathology, molecular information related to the tumor, radiology, treatment characteristics and quality of life (QoL) associated with their lymphoma care will be collected over the course of 4 years by clinical research teams at every participating institution. The de-identified data will be securely shared through a password protected REDCap with other participating institutions under data usage agreements of the consortium. Next generation sequencing (NGS) including but not limited to whole exome sequencing and bulk RNA-sequencing will be performed on archived lymphoma specimens, mononuclear cells, cfDNA and saliva (when feasible) for a comprehensive molecular characterization of the tumor. Molecular data will be analyzed in correlation with patient outcomes. Advanced deep learning algorithms will be applied to predict responses and survival across lymphoma subtypes, heterogeneous clinical scenarios and various potential therapeutic approaches that the patient has not been exposed to.

ELIGIBILITY:
Inclusion Criteria:

* Untreated, relapsed, or refractory histologically confirmed mature T-cell or NK-cell neoplasm.
* All subtypes of PTCL are eligible except for T-cell large granular lymphocytic leukemia, cutaneous T-cell lymphoma such as but not limited to mycosis fungoides and transformation, Sézary syndrome, and primary cutaneous CD30+ disorders.

Exclusion Criteria:

* Precursor T/NK neoplasms, T-cell large granular lymphocytic leukemia, cutaneous T-cell lymphoma such as but not limited to mycosis fungoides and transformation, Sézary syndrome, and primary cutaneous CD30+ disorders.
* Adults who are unable to consent, individuals who are not yet adults such as infants, children and teenagers, pregnant women, and prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational non-interventional study with the primary objective to define overall survival and time to next treatment, as well as determining the ability to bridge patients to stem cell transplantation for patients with a new diagnosis, primary refractory or relapse of T-cell or NK-cell neoplasm.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 4 Years
  Difference in overall survival (OS) in subjects with primary refractory versus relapsed mature T-cell and NK-cell neoplasms at the completion of 4 years.
Progression-free Survival | Up to 4 Years
  Difference in progression-free survival (PFS) in subjects with primary refractory versus relapsed mature T-cell and NK-cell neoplasms at the completion of 4 years.
Duration of Response | Up to 4 Years
  Difference in duration of response in subjects with mature T-cell and NK-cell neoplasms treated with cytotoxic chemotherapy versus prespecified non-chemotherapeutic choice at the completion of 4 years.
Time to progression | Up to 4 Years
  Difference in time to progression in subjects with mature T-cell and NK-cell neoplasms treated with cytotoxic chemotherapy versus prespecified non-chemotherapeutic choice at the completion of 4 years.
Number of subjects proceeding to stem cell transplantation | Up to 4 Years
  Difference in number of subjects bridged to stem cell transplantation (allogeneic or autologous) with mature T-cell and NK-cell neoplasms treated with cytotoxic chemotherapy versus prespecified non-chemotherapeutic choice at the completion of 4 years.
Association of tumor specific somatic variants with treatment response | Up to 4 Years
  Determine whether tumor specific somatic variants identified at the time of diagnosis predicts response to treatment in subjects with mature T-cell and NK-cell neoplasms at the completion of 4 years in at least 50% of the patients.

SECONDARY OUTCOMES:
Complete Response Rate | Up to 4 Years
  Difference in complete response rate in subjects with mature T-cell and NK-cell neoplasms treated with cytotoxic chemotherapy versus prespecified non-chemotherapeutic choice.
Overall Response Rate | Up to 4 Years
  Difference in overall response rate in subjects with mature T-cell and NK-cell neoplasms treated with cytotoxic chemotherapy versus prespecified non-chemotherapeutic choice.
Rate of Adverse Events | Up to 4 Years
  Frequency of adverse events in subjects with mature T-cell and NK-cell neoplasms treated with cytotoxic chemotherapy versus prespecified non-chemotherapeutic choice using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

OTHER OUTCOMES:
Estimation of overall survival | Up to 4 Years
  Feasibility of Synthetic Intervention of estimating difference in overall survival as measured by the ability to predict overall survival in subjects with mature T-cell and NK-cell neoplasms treated with cytotoxic chemotherapy versus prespecified non-chemotherapeutic choice.
FACT-Lym | Up to 4 Years
  Define overall health-related quality of life as measured by the Functional Assessment of Cancer Therapy [FACT-Lym] in in subjects with mature T-cell and NK-cell neoplasms. 5-point Likert, measures 4 domains including physical, social, emotional, and functional. Ranges from 0-168, with higher scores indicating better quality of life.
FACIT-COST | Up to 4 Years
  Characterize the association between health-related quality of life as measured by the Functional Assessment of Cancer Therapy [FACT-Lym] and poverty as measured by the Functional Assessment of Chronic Illness Therapy-Comprehensive Score for Financial Toxicity [FACIT-COST] and by the Health Leads Social Needs Screening Toolkit in subjects with mature T-cell and NK-cell neoplasms. 5-point Likert with the range of 0-44, with higher scores indicate better financial well-being.
HADS | Up to 4 Years
  Describe the prevalence of psychological distress as measured by the Hospital Anxiety and Depression Scale [HADS] in subjects with mature T-cell and NK-cell neoplasms and examine whether psychological distress is associated with disease characteristics. Ranges from 0-21, with higher scores indicating higher distress (anxiety, depression).
IES-R | Up to 4 Years
  Describe the prevalence of the Impact of Event Scale-Revised [IES-R] in subjects with mature T-cell and NK-cell neoplasms and examine whether psychological distress is associated with disease characteristics and measures subjective reaction after a traumatic event. Ranges from 0-88, with higher scores indicating likely presence of PTSD.
Household Material Hardship (HMH) | Upto 4 Years
  Define the prevalence of household material hardship as measured by the Health Leads Social Needs and examine the association between household material hardship and health-related quality of life (FACT-Lym) in subjects with mature T-cell and NK-T cell neoplasms. Measures unmet concrete needs across 5 domains - housing, utility, food, transportation, interpersonal safety. Binary: no (0) or yes (1). Yes, means a positive screen with higher scores indicate greater material hardship.
Kessler Psychological Distress Scale - K10 | Upto 4 Years
  Define the prevalence of psychological distress as measured by the Kessler-10 in subjects with mature T-cell and NK-T cell neoplasms and examine whether psychological distress is associated with disease characteristics. 5-point Likert with the range of 0-24, with higher scores suggesting serious PD (psychological distress) or higher likelihood of diagnosable mental illness.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (8):
  - City of Hope, Duarte, California
  - University of Colorado, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - OhioHealth, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Japan (2):
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki, Hyōgo
  - Kyoto University, Kyoto
- University of Cape Town, Cape Town, South Africa, South Africa